CLINICAL TRIAL: NCT04866628
Title: Comparison of Helichrysum Italicum Infusion and Helichrysum Arenarium Infusion Effects on the Components of Metabolic Syndrome in Adults
Brief Title: Clinical Trials of Two Helichrysum Infusions in Adults
Acronym: SMILJ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Primorska (Other)
Responsible Party: Principal Investigator, Zala Jenko Praznikar, Associate professor, University of Primorska
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SMILJ_Clinical
Record Dates: First submitted 2021-04-23; First posted 2021-04-30 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Hypertension; Hyperlipidemias; Inflammation; Hyperglycemia; Hypercholesterolemia; Microbial Colonization; Overweight and Obesity
Keywords: metabolic syndrome; herbal infusions; diet; microbiota
MeSH Terms: conditions — Hypertension; Hyperlipidemias; Inflammation; Hyperglycemia; Hypercholesterolemia; Communicable Diseases; Overweight; Obesity; Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Helichrysum italicum (Experimental): 1 g of milled plant material (Helichrysum italicum) immersed in hot water (200 mL, 100 °C) for 10minutes
  Interventions: Dietary Supplement: Helichrysum italicum infusion
- Helichrysum arenarium (Active Comparator): 1 g of milled plant material (Helichrysum arenarium) immersed in hot water (200 mL, 100 °C) for 10minutes
  Interventions: Dietary Supplement: Helichrysum arenarium

INTERVENTIONS:
Dietary Supplement: Helichrysum italicum infusion — Comparison of metabolic syndrome components before and after four weeks of daily consumption of Helichrysum italicum infusion.
  Arms: Helichrysum italicum
Dietary Supplement: Helichrysum arenarium — Comparison of metabolic syndrome components before and after four weeks of daily consumption of Helichrysum arenarium infusion.
  Arms: Helichrysum arenarium

SUMMARY:
The study evaluates the effects of Helichrysum italicum and Helichrysum Arenarium on different components of the metabolic syndrome. The components of metabolic syndrome will be measured at baseline and four weeks after daily consumptions of either Helichrysum italicum or either Helichrysum Arenarium, and after two weeks of washout. In addition, stool samples will be also taken at baseline and after four weeks of daily consumtion of either Helichrysum italicum or either Helichrysum Arenarium.

DETAILED DESCRIPTION:
Helichrysum arenarium (HA) has a long tradition in European ethno-medicine as a medicinal plant with many known activities; EU monograph supports its use for the digestive disorders, feeling of fullness and bloating, and, importantly, it re-ports no side effects. Assessment report of the European Medicines Agency Committee on Herbal Medicinal Products supports its stimulatory role in the bile flow and in the release of cholesterol to the bile. HA has also been used in chronic liver inflammatory disease and as a scavenger of free radicals. Similar to HA Helichrysum italicum (HI) is widely used in traditional medicine. Lately, much attention has been given to natural antioxidants and their ability to delay the progression of chronic diseases related to the formation and the activity of reactive oxygen species and other free radicals. Herbs are very often used to prepare recreational tea and are thereby important sources of antioxidants in different cultures. In traditional medicine, HI is also used in diet, mainly for the preparation of infusions in treating respiratory and digestive conditions.

Therefore,the ail of our study is to evaluate the effects of Helichrysum italicum and Helichrysum Arenarium on different components of the metabolic syndrome in adults presenting at least two components of metabolic syndrome and yet not receiving any medication. The components of metabolic syndrome (lipid profile, blood pressure, antrophometry, inflammation status, glucose levels) will be measured at baseline and four weeks after daily consumptions of either Helichrysum italicum or either Helichrysum Arenarium, and after two weeks of washout. In addition, stool samples will be also taken at baseline and after four weeks of daily consumtion of either Helichrysum italicum or either Helichrysum Arenarium.

ELIGIBILITY:
Inclusion Criteria:

* stable weight in the last 3 months
* BMI more than 25
* clinical diagnosis of at least two components of metabolic syndrome,

Exclusion Criteria:

* consumption of dietary supplements
* medications for any component of metabolic syndrome

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 30 (Actual)
Dates: Start 2021-05-06 (Actual); Primary Completion 2021-06-03 (Actual); Study Completion 2021-06-19 (Actual)

PRIMARY OUTCOMES:
Lipid profile | changes from baseline to four weeks of daily consumption and after two weeks of washout
  Changes in total cholesterol, LDL cholesterol, HDL cholesterol and triacylglycerides will be examined with biochemical analyzer Cobass

SECONDARY OUTCOMES:
Blood pressure | changes from baseline to four weeks of daily consumption and after two weeks of washout
  Systolic and diastolic blood pressure will be determined with blood pressure device (Omron M3)
Inflammation | Chages from baseline to four weeks of daily consumption and after two weeks of washout
  Changes in C-reactive protein levels will be examined with biochemical analyzer Cobass
Anthropometric measurements | Chages from baseline to four weeks of daily consumption and after two weeks of washout
  Changes in body weight (in kilograms) will be examined with bioelectrical impedance analysis (BIA) Tanita MC-980MA (Maeno-cho, Japan) and dedicated software (GMON Pro-Tanita).
Microbiota | Chages from baseline to four weeks of daily consumption and after two weeks of washout
  The microbiota composition will be determined with gene sequencing
Antioxidative potential | Chages from baseline to four weeks of daily consumption and after two weeks of washout
  Antioxidative potential will be determined with DPPH radical measuremen
Anthropometric measurements | Chages from baseline to four weeks of daily consumption and after two weeks of washout
  Changes in visceral fat rating will be examined with bioelectrical impedance analysis (BIA) Tanita MC-980MA (Maeno-cho, Japan) and dedicated software (GMON Pro-Tanita).
Anthropometric measurements Description: | Chages from baseline to four weeks of daily consumption and after two weeks of washout
  Changes in fat (percentage of body fat) will be examined with bioelectrical impedance analysis (BIA) Tanita MC-980MA (Maeno-cho, Japan) and dedicated software (GMON Pro-Tanita).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Primorska, Faculty of Health Sciences, Izola, Slovenia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Pljevljakusic D, Bigovic D, Jankovic T, Jelacic S, Savikin K. Sandy Everlasting (Helichrysum arenarium (L.) Moench): Botanical, Chemical and Biological Properties. Front Plant Sci. 2018 Aug 7;9:1123. doi: 10.3389/fpls.2018.01123. eCollection 2018. PMID 30131818
- [Background] Sala A, Recio M, Giner RM, Manez S, Tournier H, Schinella G, Rios JL. Anti-inflammatory and antioxidant properties of Helichrysum italicum. J Pharm Pharmacol. 2002 Mar;54(3):365-71. doi: 10.1211/0022357021778600. PMID 11902802
- [Background] Kramberger K, Jenko Praznikar Z, Baruca Arbeiter A, Petelin A, Bandelj D, Kenig S. A Comparative Study of the Antioxidative Effects of Helichrysum italicum and Helichrysum arenarium Infusions. Antioxidants (Basel). 2021 Mar 3;10(3):380. doi: 10.3390/antiox10030380. PMID 33802628